CLINICAL TRIAL: NCT01413061
Title: Study of Subtalar Arthrodesis Using AlloStem® Versus Autologous Bone Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AlloSource (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlloSource Subtalar Fusion RCT
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Degenerative Osteoarthritis; Post-traumatic; Arthrosis; Rheumatoid Arthritis & Other Inflammatory Polyarthropathies; Rheumatoid Arthritis of Subtalar Joint
Keywords: Other Hindfoot Conditions requiring Subtalar Arthrodesis; Post-traumatic Arthritis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AlloStem Live Cellular Allograft (Active Comparator): AlloStem is the combination of the Mesenchymal Stem Cells (MSC) derived from adipose with demineralized bone.
  Interventions: Procedure: Subtalar Arthrodesis
- Control: Autologous Bone Marrow Aspirate (Active Comparator): Autologous bone graft is recovered from the patient's own tibia or iliac crest, for transplantation in the subtalar joint.
  Interventions: Procedure: Subtalar Arthrodesis

INTERVENTIONS:
Procedure: Subtalar Arthrodesis

SUMMARY:
The purpose of this clinical trial is to evaluate the outcome of implanting AlloStem® graft with appropriate rigid internal fixation hardware as an alternative to autograft bone graft with rigid fixation in subtalar arthrodesis procedures. The primary objective of this clinical trial is to compare the overall fusion rate of the investigational to the control treatment. Fusion will be determined by clinical findings, radiographs and computed tomography (CT) of the subtalar joint 24 weeks (6 months) after the trial surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Must be diagnosed with degenerative osteoarthritis, post-traumatic arthritis, inflammatory arthritis (ie: rheumatoid arthritis) or other conditions of the hindfoot requiring subtalar arthrodesis.
2. Patients must be able to attend follow-up examinations for the duration of the trial.
3. The patient is at least 18 years of age and skeletally mature, or less than 80 years of age at the time of surgery.
4. Is willing and able to comply with the clinical trial plan and able to understand and sign the Patient Informed Consent Form.

Exclusion Criteria:

1. Younger than 18 years old or older than 80 years old.
2. Has a condition that prevents ambulation or completion of any of the trial measurements.
3. Requires fusion of additional hindfoot or ankle joints simultaneously (i.e. a pantalar, tibiotalocalcaneal or triple arthrodesis). Concomitant midfoot or forefoot procedures, such as osteotomies, tendon or metatarsal procedures are not exclusionary.
4. Has treatment planned for the arthrodesis which does not require the use of screws.
5. Has any active infection of the hindfoot, a systemic infection or bacteremia.
6. Has received any treatment within the past 12 months which may interfere with bone metabolism [bisphosphonates (Fosamax, Actonel, Boniva, Reclast) and calcitonin (Miacalcin)].
7. Is scheduled to have any surgical procedure on the contralateral foot within 6 weeks before or after the study procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Fusion Rate (%)(as determined by CT assessment) | 6 months post-op
  Fusion Rate (%)(as determined by CT assessment)

SECONDARY OUTCOMES:
Radiographic outcome assessments | Pre-operatively, 6 weeks, 3, 6, 12 and 24 months
  Radiographic outcome assessments
Functional outcome measurements | Pre-operatively, 6 weeks, 3, 6, 12 and 24 months
  FFI-R, SF-12
Functional outcome measurements | Pre-operatively, 3, 6, 12 and 24 months
  AOFAS

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Coetzee, MD, Principal Investigator — Minnesota Orthopedic Sports Medicine Institute (MOSMI); Mark Myerson, MD, Principal Investigator — Institute for Foot and Ankle Reconstruction at Mercy; John Anderson, MD, Principal Investigator — Orthopaedic Associates of Michigan; Paul Juliano, MD, Principal Investigator — Milton S. Hershey Medical Center; Andrew Murphy, MD, Principal Investigator — Campbell Clinic
Locations (5):
- United States (5):
  - Institute for Foot and Ankle Reconstruction at Mercy, Baltimore, Maryland
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Minnesota Orthopedic Sports Medicine Institute (MOSMI), Edina, Minnesota
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Campbell Clinic, Germantown, Tennessee